CLINICAL TRIAL: NCT05740865
Title: Predicting Deep Surgical Site Infection in Patients Receiving Open Posterior Instrumented Thoracolumbar Surgery--- A-DOUBLE-SSI Risk Score: a Large Retrospective Multicenter Cohort Study in China
Brief Title: Risk Factors Associated With Infection After Spine Surgery
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: Neurospine_infection
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Deep Surgical Site Infection; Spine Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who developed deep surgical site infection after thoracolumbar surgery: this group included patients who developed deep surgical site infection after open posterior instrumented thoracolumbar surgery
  Interventions: Procedure: open posterior instrumented thoracolumbar surgery
- patients who did not develop deep surgical site infection after thoracolumbar surgery: this group included patients who did not develop deep surgical site infection after open posterior instrumented thoracolumbar surgery
  Interventions: Procedure: open posterior instrumented thoracolumbar surgery

INTERVENTIONS:
Procedure: open posterior instrumented thoracolumbar surgery — Both group previously received open posterior instrumented thoracolumbar surgery in 4 centers

SUMMARY:
Surgical site infection (SSI), particularly deep SSI, is one of the most serious complications after spinal surgery. evaluating the risk of SSI and, correspondingly, prescription of prophylactic measures are extremely important to prevent SSI and avoid potentially devastating consequences. A retrospective study was conducted aiming to develop a point-based prediction model of deep surgical site infection in patients receiving open posterior instrumented thoracolumbar surgery.

DETAILED DESCRIPTION:
Data of 3,419 patients in 4 hospitals from Jan 1, 2012 to Dec 30, 2021 were retrospectively collected and were evaluated aiming to develop a point-based prediction model of deep surgical site infection in patients receiving open posterior instrumented thoracolumbar surgery. Clinical knowledge-driven, data-driven and decision tree model was used to identify predictive variables of deep SSI. Internal validation was performed by using bootstrapping methods.

ELIGIBILITY:
Inclusion Criteria:

patients who previously received open posterior instrumented thoracolumbar surgery

Exclusion Criteria:

1. were aged < 18 years;
2. underwent surgery for the spinal infection, spine revision surgery, or cervical operation;
3. were diagnosed as superficial SSI;
4. died in hospital;
5. diagnosis of SSI was not determined;
6. had missing data more than 10% were excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population included patients who previously receceived open posterior instrumented thoracolumbar surgery due to spine disease (except that spine infection or revision surgery)
Sampling Method: Non-Probability Sample
Enrollment: 3419 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
deep surgical site infection | within 30 days after the operation
  deep SSI was defined as an infection occurring within 30 days after the operation involving deep soft tissues along with one of the following criterion: (1)purulent drainage from the deep incision but not from the organ/space component of the surgical site;(2) a deep incision spontaneously dehisces or is deliberately opened by a surgeon when the patient has at least one of the following signs or symptoms: fever >38℃, localized pain, or tenderness, unless site is culture-negative;(3) an abscess or other evidence of infection involving the deep incision is found on direct examination, during reoperation, or by histopathologic or radiologic examination;(4) diagnosis of a deep incisional SSI by a surgeon or attending physician. In this study, organ space SSI was also classified as deep SSI due to the same criteria as deep SSI.

CONTACTS AND LOCATIONS:
Overall Officials: Fengzeng Jian, Study Director — Xuanwu Hospital, China International Neuroscience Institute, Capital Medical University
Locations (1):
- Xuanwu Hospital, China International Neuroscience Institute, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheng L, Liu J, Lian L, Duan W, Guan J, Wang K, Liu Z, Wang X, Wang Z, Wu H, Chen Z, Wang J, Jian F. Predicting deep surgical site infection in patients receiving open posterior instrumented thoracolumbar surgery: A-DOUBLE-SSI risk score - a large retrospective multicenter cohort study in China. Int J Surg. 2023 Aug 1;109(8):2276-2285. doi: 10.1097/JS9.0000000000000461. PMID 37204435